CLINICAL TRIAL: NCT03673293
Title: Measuring Postoperative Mobility, Gait Symmetry and Feedback With New Technology Following Total Joint Arthroplasty
Brief Title: Measuring Postoperative Mobility, Gait Symmetry and Feedback Following TJA
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Christopher Pelt, Principle Investigator, University of Utah
Other Study IDs: 110935
Record Dates: First submitted 2018-09-12; First posted 2018-09-17 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Total Joint Arthroplasty
Keywords: Total Joint Arthroplasty; Postoperative mobility; Gait symmetry; Feedback

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objectives of this study are:

1. The investigators plan to evaluate and validate the use of a novel wireless insole device (Loadsol) that provides real-time biofeedback on post-operative mobility and weight bearing following total joint arthroplasty.
2. The investigators plan to utilize the wireless insole device to determine if biofeedback is sufficient for improving gait symmetry following total joint arthroplasty.
3. The investigators plan to determine if there is a correlation between patient reported outcomes and measured postoperative weight bearing.

DETAILED DESCRIPTION:
In orthopaedic and trauma surgery post-operative mobility is very important. Six-month mortality and patient satisfaction has been associated with mobility. Elderly patients may suffer from severe complications caused by immobility due to a high prevalence of comorbidities.

Measuring postoperative mobility has primarily been based on advanced technology and complicated gait laboratories (treadmill, force plate, videoanalysis). The recent introduction of mobile insole force devices, such as the pedoped loadsol® (Novel) may allow for a cost-effective and clinically relevant use of providing biofeedback.

Using video analysis to evaluate the insole device will allow for measurements in realistic situations like walking stairs, stand up from a chair, sit down, turning and walking. The investigators had previously completed this in the lab setting and further the feedback mode of the loadsol will be used for training the patients in terms of symmetry after a total knee replacement.

This study may have an important influence on the aftercare of the investigators patients. Determining the postoperative mobility and evaluating gait analysis in real time will allow the investigators to compare between different operative approaches, operative techniques, Implants and more. If the feedback mode is working as expected the investigators might use it in the close future in the investigators standard aftercare for all patients.

ELIGIBILITY:
Inclusion Criteria:

* Planned or recently underwent (up to 8 weeks postoperatively) primary total joint arthroplasty
* Free walking before surgery, no devices needed
* Age >/=18 years
* Preoperative outcomes scores (PF CAT, PROMIS Global Health, KOOS JR)
* Written informed consent

Exclusion Criteria:

* Index procedure is a revision total joint arthroplasty
* Total knee or hip arthroplasty on the contralateral side within 1 one year of index procedure
* Severe medical comorbidity (ASA>/=3)
* Participant is planning TJA on another joint within next 12 months
* Significant symptoms on contralateral knee/hip/ankle that could impede performance on study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who plan or recently underwent (up to 8 weeks postoperatively) primary total joint arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2018-05-05 (Actual); Primary Completion 2025-08-08 (Actual); Study Completion 2025-08-08 (Actual)

PRIMARY OUTCOMES:
Peak Vertical Ground Reaction Forces (vGRF) | 6-weeks
  Gait analysis of vertical ground reaction forces generated while performing routine exercises
Peak Vertical Ground Reaction Forces (vGRF) | 6-months
  Gait analysis of vertical ground reaction forces generated while performing
Peak Vertical Ground Reaction Forces (vGRF) | 12-months
  Gait analysis of vertical ground reaction forces generated while performing

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Pelt, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Orthopaedic Center, Salt Lake City, Utah, United States